CLINICAL TRIAL: NCT05820022
Title: Evaluating Scientific Research Barriers by Gender and Other Characteristics From the Perspective of Physiatrists in Turkey: A Multicenter Survey Study
Brief Title: Scientific Research Barriers by Gender and Other Characteristics in Physiatry
Status: Completed | Type: Observational
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: Barrier1
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Gender Bias; Researcher-Subject Relations
MeSH Terms: conditions — Sexism

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physical Medicine and Rehabilitation Specialists: Physical medicine and rehabilitation specialists
  Interventions: Other: Research Barriers Scale

INTERVENTIONS:
Other: Research Barriers Scale — This scale was prepared after a detailed literature review and sent to five physiatrists for review and feedback. It consists of 21 items with Likert-type responses and two open-ended questions. It is designed to measure the barriers that individuals or groups face in conducting research. The scale includes a list of potential barriers and asks respondents to rate the extent to which they experience each barrier. Examples of barriers that may be included in such a scale could include lack of funding, limited access to resources or equipment, time constraints, difficulty finding participants or accessing data, institutional or administrative hurdles, and so on.

SUMMARY:
The ever-increasing population and life expectancy worldwide lead to a higher prevalence of physical disabilities and diseases, which increases the need for physical medicine and rehabilitation research. In our study, we aimed to evaluate various aspects of the barriers, particularly gender disparities, faced by physical medicine and rehabilitation professionals who wish to conduct scientific research.

DETAILED DESCRIPTION:
Physicians in physical medicine and rehabilitation must also put in tremendous effort and manage their time meticulously to contribute to scientific research (SR). Research requires knowledge, experience, and institutional support, such as financial incentives, technical facilities, and trained personnel. In this field, research productivity is increasingly important due to the rising prevalence of conditions such as age-related disability and chronic pain, which put pressure on the healthcare system and affect people's quality of life. Turkey's publication productivity in physical medicine and rehabilitation has also increased steadily in recent years, with a significant number of articles published between 2015 and 2020. However, gender disparities in academic leadership positions persist in this field as well, with women lagging behind men in the number of scientific publications. While bibliometric studies are useful for assessing the current state of scientific performance, survey studies are necessary to identify obstacles that deter researchers and increase research productivity. Unfortunately, few studies have used this approach in physical medicine and rehabilitation, and no such study has been conducted in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Being a physical medicine and rehabilitation physician.
* Giving consent to participate in the study.

Exclusion Criteria:

- Not giving consent to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physical medicine and rehabilitation physicians who consented to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Research Barriers Scale | 1 day
  This scale was prepared after a detailed literature review and sent to five physiatrists for review and feedback. It consists of 21 items with Likert-type responses and two open-ended questions. It is designed to measure the barriers that individuals or groups face in conducting research. The scale includes a list of potential barriers and asks respondents to rate the extent to which they experience each barrier. Examples of barriers that may be included in such a scale could include lack of funding, limited access to resources or equipment, time constraints, difficulty finding participants or accessing data, institutional or administrative hurdles, and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital
Locations (1):
- Üsküdar State Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon reasonable request by the principal investigator.